CLINICAL TRIAL: NCT03152903
Title: A Multicenter Phase II/III Double-Blind, Randomized, Placebo Controlled Study To Evaluate The Efficacy And Safety Of VPM1002 In The Prevention Of Tuberculosis (TB) Recurrence In Pulmonary TB Patients After Successful TB Treatment
Brief Title: Study to Check the Efficacy and Safety of Recombinant BCG Vaccine in Prevention of TB Recurrence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VPM1002-IN-3.01TBR
Record Dates: First submitted 2017-04-28; First posted 2017-05-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Prevention of TB Recurrence
Keywords: Recombinant BCG vaccine; Category 1 pulmonary tuberculosis; Recurrence; Efficacy
MeSH Terms: conditions — Recurrence | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VPM1002 (Recombinant BCG vaccine) (Experimental)
  Interventions: Biological: VPM1002 (Recombinant BCG Vaccine)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VPM1002 (Recombinant BCG Vaccine) — VPM1002 is a formulated, lyophilized cake of live recombinant Mycobacterium bovis rBCGÄureC::Hly+; VPM1002.
  VPM1002 is the active pharmaceutical ingredient. It is a genetically modified BCG vaccine derived from the Mycobacterium bovis BCG subtype Prague characterized as rBCGÄureC::Hly+. Single dose of VPM1002 is administered intradermally.
  Arms: VPM1002 (Recombinant BCG vaccine)
Other: Placebo — Single dose of Placebo is administered intradermally.
  Arms: Placebo

SUMMARY:
This is a Phase II/III trial with two groups of adults successfully cured of category 1 pulmonary TB receiving either VPM1002 or placebo. Single dose of VPM1002 / placebo will be administered to calculate efficacy of the vaccine against TB recurrence.

DETAILED DESCRIPTION:
The study is designed as a multicenter, double-blinded, randomized, placebo-controlled trial with two groups of category 1 pulmonary TB patients who have successfully completed ATT and declared cured by bacteriological confirmation.

The eligible participants will be randomized in 1:1 ratio to receive single dose of either VPM1002 or placebo. After study vaccination, participants will be followed up for one year. Any suspected TB case during follow up will be further evaluated and bacteriologically confirmed. Study participants will be actively followed up for 2 months post-vaccination for any solicited local and regional reaction. SAEs will be recorded and reported throughout study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18 and ≤65 years.
2. Bacteriologically confirmed Category I pulmonary TB patients (including controlled diabetics with HbA1c level ≤7% and non-diabetics) who successfully completed ATT as per national guidelines.
3. Must have a sputum sample showing bacteriologic confirmation of cure - defined as smear negative.
4. Female participants who are currently using reliable methods of birth control, have a negative pregnancy test during screening and have no intention to become pregnant for at least 3 months post-vaccination.
5. Participant must intend to remain in the area during the study period.

Exclusion Criteria:

1. Reactive serology for HIV
2. History of extrapulmonary TB
3. Known or suspected impairment of immunological function
4. Pregnant and / or lactating female participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Percentage of bacteriologically confirmed TB recurrence cases | 2-12 months post-vaccination
  Percentage of TB recurrence patients who have previously been successfully treated for TB, were declared cure and are now diagnosed with a new episode of bacteriologically confirmed recurrent TB after at least 2 months from vaccination.

SECONDARY OUTCOMES:
Percentage of overall TB recurrence (i.e. either bacteriologically confirmed or clinically diagnosed TB recurrence) | 2-12 months post-vaccination
  Percentage of TB recurrence patients who have previously been successfully treated by for TB, were declared cure and are now diagnosed with a new episode of either bacteriologically confirmed or clinically diagnosed recurrent TB after at least 2 months from vaccination.
Safety assessed by Solicited local and regional reactogenicity and Unsolicited adverse events and SAEs | Throughout study participation i.e.12 months post-vaccination
  * Solicited local and regional reactogenicity events within 2 months following study vaccination
  * Unsolicited adverse events and SAEs throughout the study period

CONTACTS AND LOCATIONS:
Locations (10):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh
- India (9):
  - Mahavir Hospital & Research Centre, Hyderabad, Hyderabad, Andhra Pradesh
  - Government Medical College, Jammu, Jammu, Jammu and Kashmir
  - B.J. Govt. Medical College and Sassoon General Hospitals, Pune, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Sevagram, Sevāgrām, Maharashtra
  - Christian Medical College and Hospital, Ludhiana, Ludhiana, Punjab
  - MV Hopsital for Diabetes Pvt Ltd, Chennai, Chennai, Tamil Nadu
  - Sri Ramachandra Hospital Chennai, Chennai, Tamil Nadu
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry, Tamil Nadu
  - Christian Medical College and Hospital, Vellore, Vellore, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giersing B, Mo AX, Hwang A, Baqar S, Earle K, Ford A, Deal C, Dull P, Friede M, Hall BF. Meeting summary: Global vaccine and immunization research forum, 2023. Vaccine. 2025 Feb 6;46:126686. doi: 10.1016/j.vaccine.2024.126686. Epub 2025 Jan 5. PMID 39752894